CLINICAL TRIAL: NCT06292780
Title: A Phase 1/2 Study of Linvoseltamab in Patients With Relapsed or Refractory Systemic Light Chain Amyloidosis
Brief Title: A Trial to Learn if Linvoseltamab is Safe and Works in Adults With Relapsed or Refractory Systemic Light Chain Amyloidosis (AL Amyloidosis)
Acronym: LINKER-AL2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-2274; 2023-507809-34-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-03

CONDITIONS: Relapsed/Refractory Systemic Light Chain Amyloidosis
Keywords: Amyloid light-chain (AL); Multiple Myeloma (MM); Pathogenic light chains
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Note: Participants enrolled in Phase 2 will be randomized 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Cohort 1: Low Dose (Experimental): Dose Escalation: Non-Randomized
  Interventions: Drug: Linvoseltamab
- Phase 1: Cohort 2: High Dose (Experimental): Dose Escalation: Non-Randomized
  Interventions: Drug: Linvoseltamab
- Phase 2: Low Dose (Experimental): Dose Expansion: Participants will be randomized in a 1:1 ratio
  Interventions: Drug: Linvoseltamab
- Phase 2: High Dose (Experimental): Dose Expansion: Participants will be randomized in a 1:1 ratio
  Interventions: Drug: Linvoseltamab

INTERVENTIONS:
Drug: Linvoseltamab — anti-B-cell maturation antigen x anti-Cluster of differentiation 3 bispecific antibody
  Other Names: REGN5458; Lynozyfic™

SUMMARY:
This study is researching an experimental drug called linvoseltamab ("study drug").

This study is focused on patients who have AL amyloidosis that has returned or have failed other therapies and need to be treated again.

The study consists of 2 phases (Phase 1 and Phase 2):

* In Phase 1, linvoseltamab will be given to a small number of participants to study the side effects of the study drug and to determine the recommended doses of the study drug to be given to participants in Phase 2.
* In Phase 2, linvoseltamab will be given to more participants to continue to assess the side effects of the study drug and to evaluate the ability of linvoseltamab to treat AL amyloidosis.

The study is looking at several other research questions, including:

* How many participants treated with linvoseltamab have improvement in the abnormal proteins that cause organ problems and for how long
* How many participants treated with linvoseltamab have improvement in the heart or kidney and for how long
* What the right dosing regimen is for linvoseltamab
* What side effects may happen from taking linvoseltamab
* How much linvoseltamab is in the blood at different times
* Whether the body makes antibodies against linvoseltamab (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis of AL amyloidosis, as described in the protocol
2. Measurable disease as defined by serum difference between involved and uninvolved free light chains (dFLC) concentration, as described in the protocol
3. Previously treated after at least 1 prior therapy and requiring further treatment as assessed by the Investigator
4. N-terminal pro b-type natriuretic peptide (NT-proBNP) ≤8500 ng/L during screening
5. Adequate hepatic, hematologic, renal, and cardiac function, as described in the protocol
6. Eastern Cooperative Oncology Group (ECOG) performance score ≤2 at screening

Key Exclusion Criteria:

1. History of other non-AL amyloidosis
2. Greater than 60% plasmacytosis on a bone marrow biopsy and/or aspirate during screening
3. Presence of lytic bone lesion(s) or extramedullary plasmacytoma on imaging during screening
4. Myocardial infarction within the past 6 months prior to the first screening visit
5. Known active infection requiring hospitalization or treatment with IV anti-infectives within 28 days of first administration of study drug

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2028-08-20 (Estimated); Study Completion 2035-02-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLTs) | Up to 28 Days
  Phase 1
Achievement of hematologic complete response (CR) as determined by the Independent Review Committee (IRC) | Up to 3 years
  Phase 2

SECONDARY OUTCOMES:
Achievement of hematologic CR, as determined by the IRC | Up to 3 years
  Phase 1
Achievement of hematologic very good partial response (VGPR) or better response (CR + VGPR), as determined by the IRC | Up to 3 years
Achievement of overall hematologic response (PR or better), as determined by the IRC | Up to 3 years
Time to initial hematologic response | Up to 3 years
Time to best hematologic response | Up to 3 years
Duration of hematologic response (ie, best response, VGPR or better, overall response), as determined by the IRC | Up to 7 years
Hematologic progression-free survival (PFS) | Up to 7 years
Incidence of death | Up to 7 years
Incidence of treatment-emergent adverse events (TEAEs) | Up to 39 months
Severity of TEAEs | Up to 39 months
Incidence of serious adverse events (SAEs) | Up to 39 months
Severity of SAEs | Up to 39 months
Incidence of adverse events of special interest (AESIs) | Up to 39 months
Severity of AESIs | Up to 39 months
Achievement of overall hematologic response (PR or better), as determined by the IRC in dose regimen 1 vs 2 | Up to 39 months
  Phase 2
Incidence of TEAEs in dose regimen 1 vs 2 | Up to 39 months
  Phase 2
Severity of TEAEs in dose regimen 1 vs 2 | Up to 39 months
  Phase 2
Incidence of SAEs in dose regimen 1 vs 2 | Up to 39 months
  Phase 2
Severity of SAEs in dose regimen 1 vs 2 | Up to 39 months
  Phase 2
Incidence of AESIs in dose regimen 1 vs 2 | Up to 39 months
  Phase 2
Severity of AESIs in dose regimen 1 vs 2 | Up to 39 months
  Phase 2
Time from treatment initiation to hematologic disease progression as determined by the IRC | Up to 7 years
Time from treatment initiation to cardiac deterioration, as determined by the IRC | Up to 7 years
Time from treatment initiation to kidney deterioration as determined by the IRC | Up to 7 years
Time from treatment initiation to death as determined by the IRC | Up to 7 years
Time from initiation of treatment to date of death from any cause | Up to 7 years
Achievement of renal response in participants with renal involvement at baseline, as determined by IRC | Up to 7 years
Achievement of cardiac response in participants with cardiac involvement at baseline, as determined by IRC | Up to 7 years
Time to first renal response in participants with renal involvement at baseline | Up to 7 years
Time to first cardiac response in participants with cardiac involvement at baseline | Up to 7 years
Linvoseltamab concentration in serum over time | Up to 39 months
Incidence of anti-drug antibodies (ADAs) to linvoseltamab over time | Up to 39 months
Titers of ADAs to linvoseltamab over time | Up to 39 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (18):
- United States (7):
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute/SCRI, Denver, Colorado
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Ohio State University, Columbus, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital - The Catholic University of Korea, Seoul
- Spain (5):
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Hospital de Cabuenes, Gijón, Principality of Asturias
  - Universität de Barcelona- Institut d' Investigacions Biomediques August Pi i Sunyer (IDIBAPS), Barcelona
  - University Hospital La Fe, Valencia
- United Kingdom (2):
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/